CLINICAL TRIAL: NCT05731154
Title: Development of an Artificial Intelligence Solution to Evaluate Clinical Activity of Thyroid Associated Orbitopathy Using Periocular Selfie Images Taken by Smartphones in Patients With Thyroid Dysfunction
Brief Title: Development of an AI Solution to Evaluate Clinical Activity of TAO Using Periocular Images Taken by Smartphones in Patients With Thyroid Dysfunction
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: THYROSCOPE INC. (Industry)
Responsible Party: Principal Investigator, Namju Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-2110-715-304
Record Dates: First submitted 2022-04-17; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Thyroid Eye Disease
Keywords: thyroid eye disease; artificial intelligence; machine learning; smartphone
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- thyroid eye disease group: Patients who were diagnosed as thyroid eye disease. Periorbital images are taken by DSLR camera in the studio. Periorbital selfie images are taken by the patients with 6 smartphones including various camera modules.
  CAS of TAO is evaluated by 3 ophthalmologists based on the periorbital digital images taken by DSLR camera and symptoms.
  Interventions: Other: taking periorbital selfie images using smartphones

INTERVENTIONS:
Other: taking periorbital selfie images using smartphones — taking periorbital selfie images using smartphones

SUMMARY:
This study was conducted to develop an AI solution to evaluate clinical activity score (CAS) of thyroid associated orbitopathy (TAO) using periocular selfie images taken by smartphones in patients with thyroid dysfunction.

An AI solution to evaluate CAS in TAO was developed in previous retrospective study using periorbital digital images taken by DSLR camera in the studio. This AI solution will be adjusted to show its best performance with periocular selfie images taken by smartphones.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thyroid eye disease

Exclusion Criteria:

* Patients who have prior facial anomaly or surgery
* Patients who cannot use smartphone camera app

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is conducted to develop AI solution using smartphone selfie images. Therefore, the number of subjects for this study was calculated as 200, the maximum number of patients with thyroid eye disease that can be prospectively recruited during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Accuracy for clinical activity score (CAS) of thyroid eye disease (TED) | baseline (this study has no intervention)
  Accuracy of AI solution using smartphone selfie images for CAS of TED.
Diagnostic accuracy for active thyroid eye disease | baseline (this study has no intervention)
  Accuracy of AI solution using smartphone selfie images for active thyroid eye disease (TED) which is defined as 3 or more of clinical activity score

SECONDARY OUTCOMES:
Accuracy for redness of eyelids | baseline (this study has no intervention)
  Accuracy of AI solution using smartphone selfie images for redness of eyelids
Accuracy for redness of conjunctiva | baseline (this study has no intervention)
  Accuracy of AI solution using smartphone selfie images for redness of conjunctiva
Accuracy for swelling of eyelids | baseline (this study has no intervention)
  Accuracy of AI solution using smartphone selfie images for swelling of eyelids
Accuracy for swelling of conjunctiva | baseline (this study has no intervention)
  Accuracy of AI solution using smartphone selfie images for swelling of conjunctiva
Accuracy for swelling of caruncle | baseline (this study has no intervention)
  Accuracy of AI solution using smartphone selfie images for swelling of caruncle

CONTACTS AND LOCATIONS:
Overall Officials: Namju Kim, MD, PhD., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.